CLINICAL TRIAL: NCT06823570
Title: Anti-hypertensive Therapy and Exercise Treatment to Improve Vascular Health in Patients With Hypertension. A Randomized Controlled Trial.
Brief Title: Anti-hypertensive Therapy and Exercise Treatment to Improve Vascular Health in Patients With Hypertension.
Acronym: Antitension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-2603
Record Dates: First submitted 2025-02-03; First posted 2025-02-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Hypertension; Vascular Function; Fitness Testing; Metabolism Changes
Keywords: cardiorespiratory fitness; retinal microcirculation; endothelial function; exercise training; lifestyle treatment
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualized exercise training group (Active Comparator): Beside a guideline based anti-hypertensive therapy, patients in the intervention group will receive an individualized exercise training program 3x/week. Exercise training will be a combination of aerobic and resistance training and is based on each patient's individual fitness level. Regular contact between exercise physiologists and patients, as well as group sessions, will help patients to maintain a regular exercise program.
  Interventions: Behavioral: Individualized exercise therapy; Behavioral: Lifestyle recommendations
- Control group (Other): Beside a guideline based anti-hypertensive therapy, patients in the lifestyle recommendation group will receive general recommendations such as salt reduction, higher physical activity levels and stress reduction.
  Interventions: Behavioral: Lifestyle recommendations

INTERVENTIONS:
Behavioral: Individualized exercise therapy — Patients in the intervention group will receive an individualized exercise training program 3x/week.
  Arms: Individualized exercise training group
Behavioral: Lifestyle recommendations — The lifestyle recommendation group will receive general recommendations such as salt reduction, higher physical activity levels and stress reduction.

SUMMARY:
This is a prospective, monocentric, randomized controlled trial to investigate the effect of anti-hypertensive treatment and/or individualized exercise training intervention on blood pressure and vascular health. Furthermore the investigators want to decipher mechanisms, which contribute to vascular health by analyzing changes in metabolism and cell function in relation to vascular reaction.

DETAILED DESCRIPTION:
Arterial hypertension is a global health burden that affects the structure and function of large and small blood vessels and induces disease-specific end-organ damage. Exercise therapy is highly recommended in the treatment of arterial hypertension to reduce blood pressure and ameliorate hypertension-induced vascular damage. Previous exercise intervention studies have shown that exercise treatment improves vascular dysfunction independently of changes in blood pressure. Several sensitive vascular biomarkers exist that could optimize risk stratification and therapeutic decisions based on the progression of individual vascular damage in patients with arterial hypertension. However, individualized vascular assessment during anti-hypertensive treatment is not yet part of routine clinical practice. In order to improve clinical decision making from a personalized medicine perspective, it is essential to better understand which vascular biomarkers have the best sensitivity in detecting therapy-induced vascular adaptations and whether anti-hypertensive therapy with or without additional exercise improves vascular health in patients with hypertension. The proposed study will evaluate the effects of guideline-directed anti-hypertensive therapy with or without individualized exercise training intervention in 60 patients with hypertension and no previous medical treatment for one year. Regular outpatient assessments of blood pressure and large and small blood vessels will be performed every two months. Anti-hypertensive therapy will be based on the current guidelines of the European Society of Hypertension. The investigators aim to achieve the target blood pressure after six months of treatment. A further six-month follow-up is planned to assess the long-term effects of anti-hypertensive therapy, with or without additional individualized exercise training intervention, on blood pressure and macro- and microvascular health. In addition, the investigators will investigate the effect of metabolic changes induced by anti-hypertensive treatment or individualized exercise training intervention on vascular health.

ELIGIBILITY:
Inclusion Criteria:

- systolic hypertension grade I-II (BP values >140 mmHg to <180 mmHg) without anti-hypertensive medication treatment

Exclusion Criteria:

* no written informed consent
* age <18 years
* isolated diastolic hypertension
* medical contraindications for the exercise treatment (for example orthopedic problems or an abnormal ECG during the cardio respiratory exercise test)
* chronic eye diseases on both eyes (for example macular degeneration or glaucoma) or high intraocular pressure (>20 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The additional effect of an anti-hypertensive treatment plus an individualizes exercise therapy on the retinal vessel diameters compared to a guideline based anti-hypertensive treatment with general lifestyle recommendations. | From enrollment to the end of treatment after six month.
  The retinal vessel diameters will be analyzed based on the arteriolar-to-venular diameter ratio (AVR).
Effect of an guideline based anti-hypertensive therapy on the retinal vessel diameters. | From enrollment to the end of treatment after six month.
  Changes of retinal vessel diameters will be analyzed based on the arteriolar-to-venular diameter ratio (AVR).

SECONDARY OUTCOMES:
The additional effect of an anti-hypertensive treatment plus an individualizes exercise therapy on the systolic and diastolic blood pressure compared to a guideline based anti-hypertensive treatment with general lifestyle recommendations. | From enrollment to the end of treatment after six month.
  Changes in unattended systolic and diastolic blood pressure in mm Hg.
Effect of an guideline based anti-hypertensive therapy on the systolic and diastolic blood pressure. | From enrollment to the end of treatment after six month.
  Changes in unattended systolic and diastolic blood pressure in mm Hg.
The additional effect of an anti-hypertensive treatment plus an individualizes exercise therapy on the microvascular endothelial function compared to a guideline based anti-hypertensive treatment with general lifestyle recommendations. | From enrollment to the end of treatment after six month.
  Changes in microvascular endothelial function will be analyzed by retinal arteriolar and venular flicker light-induced dilation.
Effect of an guideline based anti-hypertensive therapy on the microvascular endothelial function. | From enrollment to the end of treatment after six month.
  Changes in microvascular endothelial function will be analyzed by retinal arteriolar and venular flicker light-induced dilation.
The additional effect of an anti-hypertensive treatment plus an individualizes exercise therapy on the arterial stiffness compared to a guideline based anti-hypertensive treatment with general lifestyle recommendations. | From enrollment to the end of treatment after six month.
  Changes in arterial stiffness will be analyzed based on the central pulse wave velocity.
Effect of an guideline based anti-hypertensive therapy on arterial stiffness. | From enrollment to the end of treatment after six month.
  Changes in arterial stiffness will be analyzed based on the central pulse wave velocity.
The additional effect of an anti-hypertensive treatment plus an individualizes exercise therapy on physical fitness compared to a guideline based anti-hypertensive treatment with general lifestyle recommendations. | From enrollment to the end of treatment after six month.
  Changes of physical fitness will be analyzed based on cardiopulmonary exercise tests to evaluate peak oxygen uptake (VO2peak).
Effect of an guideline based anti-hypertensive therapy on physical fitness. | From enrollment to the end of treatment after six month.
  Changes of physical fitness will be analyzed based on cardiopulmonary exercise tests to evaluate peak oxygen uptake (VO2peak).
The additional effect of an anti-hypertensive treatment plus an individualizes exercise therapy on the NO metabolism of stored blood samples compared to a guideline based anti-hypertensive treatment with general lifestyle recommendations. | From enrollment to the end of treatment after six month.
  Changes of the NO metabolism will be analyzed based on nitrite, nitrate, ADMA and SDMA with nuclear magnetic resonance spectroscopy and established ELISA kits based on collected and stored blood samples.
Effect of a guideline based anti-hypertensive therapy on the NO metabolism of stored blood samples. | From enrollment to the end of treatment after six month.
  Changes of the NO metabolism will be analyzed based on nitrite, nitrate, ADMA and SDMA with nuclear magnetic resonance spectroscopy and established ELISA kits based on collected and stored blood samples.
The additional effect of an anti-hypertensive treatment plus an individualizes exercise therapy on the metabolic profile of stored blood samples compared to a guideline based anti-hypertensive treatment with general lifestyle recommendations. | From enrollment to the end of treatment after six month.
  Changes of the metabolic profile of stored blood samples will be analyzed by liquid chromatography and high-resolution tandem mass spectrometry.
Effect of a guideline based anti-hypertensive therapy on the metabolic profile of stored blood samples. | From enrollment to the end of treatment after six month.
  Changes of the metabolic profile of stored blood samples will be analyzed by liquid chromatography and high-resolution tandem mass spectrometry.
The additional effect of an anti-hypertensive treatment plus an individualizes exercise therapy on systemic inflammation markers compared to a guideline based anti-hypertensive treatment with general lifestyle recommendations. | From enrollment to the end of treatment after six month.
  Changes of systemic inflammation markers, such as cytokines, will be analyzed by ELISA and OLINK based on stored blood samples.
Effect of a guideline based anti-hypertensive therapy on systemic inflammation markers of stored blood samples. | From enrollment to the end of treatment after six month.
  Changes of systemic inflammation markers, such as cytokines, will be analyzed by ELISA and OLINK based on stored blood samples.

OTHER OUTCOMES:
The additional effect of an anti-hypertensive treatment plus an individualizes exercise therapy on fat and muscle mass compared to a guideline based anti-hypertensive treatment with general lifestyle recommendations. | From enrollment to the end of treatment after six month.
  Changes in fat and muscle mass will be investigated by bioimpedance analysis.
Effect of a guideline based anti-hypertensive therapy on fat and muscle mass. | From enrollment to the end of treatment after six month.
  Changes in fat and muscle mass will be investigated by bioimpedance analysis.
The additional effect of an anti-hypertensive treatment plus an individualizes exercise therapy on intra- and extracellular water volume compared to a guideline based anti-hypertensive treatment with general lifestyle recommendations. | From enrollment to the end of treatment after six month.
  Changes in intra- and extracellular water volume will be investigated by bioimpedance analysis.
Effect of a guideline based anti-hypertensive therapy on intra- and extracellular water volume. | From enrollment to the end of treatment after six month.
  Changes in intra- and extracellular water volume will be investigated by bioimpedance analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik Düsseldorf, Düsseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, selected study data will be shared.